CLINICAL TRIAL: NCT06710054
Title: Recording Cyclist Crashes and Long-term Injury Consequences by New Smart Tools
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Odd Mjåland, Principal investigator, Sorlandet Hospital HF
Other Study IDs: ReCyclist
Record Dates: First submitted 2022-05-19; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2022-06

CONDITIONS: Brief Description of the Focus of the Study: Number of Injuries to Bicyclists and Micro Mobility Users
Keywords: bicyclist injuries bicyclist accidents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Recording Cyclist Crashes and Long-term Injury Consequences by new Smart Tools

DETAILED DESCRIPTION:
The ReCyCLIST project is a collaboration between research institutes from the health and transport sciences, public authorities, medical expertise and web-tool developers, and end-user organisations, and as such an excellent example of a project that promotes and supports cooperation between research groups and users of the research.

Three major research questions are addressed in the ReCyCLIST project:

1. What are the numbers, characteristics and locations of accidents and injuries among cyclists and e-scooter/micro mobility device users in a representative county (Agder) in Norway?
2. What are the consequences of injuries in terms of social and individual costs including long-term consequences with respect to recovery, disability rates etc.?
3. What are the overall health impacts of cycling, when including the more comprehensive set of positive and negative effects; and what are the economic impacts from increased cycling (in terms of cost-benefit ratios)? To answer these research questions, the investigators will develop a new digital registration tool to record accidents and injuries among cyclists and users of micro mobility devices in Agder county in Norway. Patients will be followed up and data on medical rehabilitation, recovery and general conditions will be collected by use of questionnaires after three and twelve months. To map long-term consequences of injuries (> 1 year), a retrospective study will be applied based on linking data from different registers containing information about health, welfare benefits and injuries.

ELIGIBILITY:
Inclusion Criteria:

* All cyclist (including micromobility devices), with recent accidents submitted to out- and in patient clinics in a well defined region of 310 000 inhabitants

Exclusion Criteria:

* No informed consent
* "Patients" not eligible for follow up within our region

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cyclists with recent accident in our well defined region
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Time to recover | From the inclusion of bicycle accidents to 12 months after the inclusion
  Time to recover

CONTACTS AND LOCATIONS:
Locations (1):
- Sorlandet Hospital, Kristiansand, Norway